CLINICAL TRIAL: NCT06728124
Title: A Multicenter, Randomized, Double-Blind, Parallel, Placebo-Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of GZR18 Injection in Adult Obese/Overweight Subjects
Brief Title: A Phase III Clinical Study to Evaluate the Efficacy and Safety of GZR18 Injection in Adult Obese/Overweight Subjects
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GZR18-BWM-301
Record Dates: First submitted 2024-12-05; First posted 2024-12-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2024-12

CONDITIONS: Obesity/Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GZR18 (Experimental)
  Interventions: Drug: GZR18
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GZR18 — Used as specified in the protocol
  Arms: GZR18
Other: Placebo — Administered the same volume as GZR18
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase III clinical study in adult obese/overweight subjects in China to evaluate the efficacy and safety of GZR18 Injection in the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (as of the date of signing the Informed Consent Form (ICF)), male or female.
* Obese (BMI ≥ 28 kg/m2) or overweight (24 kg/m2 ≤ BMI < 28 kg/m2) with at least one comorbidity.
* Able to understand the procedures and methods in this study; willing and able to maintain a stable diet and exercise lifestyle during the research period, and willing to sign the ICF voluntarily.
* Subjects of childbearing potential with no birth plan from the signing of ICF to 8 weeks after the last dose, willingness to take effective contraceptive measures, and no plan for sperm donation. Females of childbearing potential must not be lactating and must have negative results of pregnancy tests at screening and Visit 2 (before randomization).

Exclusion Criteria:

* Known or suspected hypersensitivity to glucagon like peptide-1 receptor agonist (GLP-1RA) drugs or excipients.
* History of drug abuse prior to screening.
* History of alcohol abuse within 6 months before screening.
* Weight change of > 5.0% within 3 months before screening (self-report).
* Presence of limb deformity or mutilation affecting height measurement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percent change in weight from baseline (%) | From Week 0 to Week 48

SECONDARY OUTCOMES:
Proportion of subjects with ≥ 10%, 15%, 20%, and 25% decrease in weight from baseline | From Week 0 to Week 48
Changes from baseline in weight | From Week 0 to Week 48
Changes from baseline in body mass index (BMI) | From Week 0 to Week 48
  weight and height will be combined to report BMI in kg/m^2
Changes from baseline in hip circumference | From Week 0 to Week 48
Changes from baseline in waist circumference | From Week 0 to Week 48
Changes from baseline in waist-hip ratio (waist circumference/hip circumference) | From Week 0 to Week 48
Treatment emergent adverse events (TEAEs) | From Week 0 to Week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, Beijing, China